CLINICAL TRIAL: NCT03763747
Title: Scoreflex NC - Scoring PTCA Catheter: A Prospective, Open Label, Multi-center, Single Arm, Observational Study Designed to Evaluate the Safety and Device Procedural Success of the Scoreflex NC Scoring PTCA Catheter in Subjects With Stenotic Coronary Arteries During Percutaneous Coronary Intervention.
Brief Title: Scoreflex NC - Scoring PTCA Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrbusNeich (Industry)
Collaborators: ClinLogix. LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-0730
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Results first posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Cardiovascular Diseases
Keywords: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Cardiovascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Scoreflex NC Scoring PTCA Catheter (Experimental): Single arm with investigational Scoreflex NC Scoring PTCA catheters
  Interventions: Device: Scoreflex NC Scoring PTCA catheter

INTERVENTIONS:
Device: Scoreflex NC Scoring PTCA catheter — To dilate coronary arteries during the subject's index procedure with Scoreflex NC Scoring PTCA catheters

SUMMARY:
A prospective, open label, multi-center, single arm, observational study designed to evaluate the acute safety and device procedural success of the Scoreflex NC Scoring Percutaneous Transluminal Coronary Angioplasty (PTCA) catheters in subjects with stenotic coronary arteries during percutaneous coronary intervention.

Two-hundred (200) subjects will be treated at up to 15 U.S. sites with the Scoreflex NC Scoring PTCA catheter during their index procedure. All subjects will be screened according to the protocol inclusion and exclusion criteria and will be followed through hospital discharge.

ELIGIBILITY:
Clinical Inclusion Criteria

1. Subject is ≥ 18 years of age.
2. Subject or a legally authorized representative must provide written informed consent prior to any study related procedures.
3. Subject must agree not to participate in any other clinical study during hospitalization for the index procedure that would interfere with the endpoints of this study.
4. Subjects must have a single or double vessel coronary artery disease (CAD) and clinical evidence of ischemic heart disease, such as CAD, stable / unstable angina or silent ischemia.

   Angiographic Inclusion Criteria
5. Subject must have de novo or restenotic lesion(s) in native coronary arteries, including in-stent restenosis suitable for percutaneous coronary intervention.
6. A maximum of two lesions, including at least one target lesion, in up to two coronary arteries.
7. Target lesion must have a reference vessel diameter (RVD) between 1.75 and 4.0 mm by visual estimation.
8. Target lesion(s) must have a diameter stenosis of ≥70% by visual estimation and may include chronic total occlusions (CTO).
9. The non-target lesion must be located in different coronary artery from the Target lesion.
10. Treatment of non-target lesion, if any, must be completed prior to treatment of target lesion and must be deemed a clinical angiographic success as visually assessed by the physician.

Clinical Exclusion Criteria:

1. Subject with a known hypersensitivity or contraindication to aspirin, heparin, bivalirudin, anti-platelet medications, or sensitivity to contrast media which cannot be adequately pre-medicated.
2. Subject with known diagnosis of STEMI or NSTEMI at index presentation or within 7 days of study screening.
3. Subject with known pregnancy or is nursing. Women of child-bearing potential should have a documented negative pregnancy test within 7 days before index procedure.
4. Planned or actual target lesion treatment with an unapproved device, atherectomy, laser, cutting balloon or thrombectomy during the index procedure.
5. A serum creatinine level > 2.0 mg/dl within 7 days prior to index procedure.
6. Cerebrovascular accident (CVA) within the past 6 months.
7. Active peptic ulcer or active gastrointestinal (GI) bleeding within the past 6 months.
8. Subject has a known left ventricular ejection fraction (LVEF) <30% (LVEF may be obtained at the time of the index procedure if the value is unknown, if necessary)
9. Target lesion located within an arterial or saphenous vein graft or graft anastomosis

   Angiographic Exclusion Criteria
10. More than two lesions requiring treatment.
11. Target lesion longer than 30 mm by visual estimation.
12. Extreme angulation (90º or greater) proximal to or within the target lesion.
13. Previous percutaneous intervention of lesions in a target vessel (including side branches) conducted within 9 months before the study procedure and located within 10 mm from the current target lesion.
14. Target lesion demonstrating severe dissection prior to planned deployment of the Scoreflex NC device
15. Unprotected left main coronary artery disease. (Greater than 50% diameter stenosis)
16. Coronary artery spasm of the target vessel in the absence of a significant stenosis.
17. Target lesion with angiographic presence of probable or definite thrombus.
18. Target lesion involves a bifurcation requiring treatment with more than one stent or pre-dilatation of a side branch >2.0 mm in diameter.
19. Non-target lesion to be treated during the index procedure meets any of the following criteria:

    * Located within a bypass graft (venous or arterial)
    * Left main location
    * Chronic total occlusion
    * Involves a bifurcation (e.g., bifurcations requiring treatment with more than 1 stent)
    * Treatment not deemed a clinical angiographic success

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, MD, Principal Investigator — Piedmont Heart Institute
Locations (9):
- United States (9):
  - The Cardiac and Vascular Institute Research Foundation, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Atlanta VA Healthcare System, Decatur, Georgia
  - Delmarva Heart Research Foundation Inc./Peninsula Regional Medical Center, Salisbury, Maryland
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - The Lindner Research Center/The Christ Hospital Heart and Vascular, Cincinnati, Ohio

REFERENCES:
- [Result] Kandzari D, Hearne S, Kumar G, Sachdeva R, Adams G, Blossom B, Dahle T, Sanghvi K, Cohen MG, Imperi G, Riley R, Almonacid AP. Procedural Effectiveness With a Focused Force Scoring Angioplasty Catheter: Procedural and Clinical Outcomes From the Scoreflex NC Trial. Cardiovasc Revasc Med. 2022 Feb;35:85-90. doi: 10.1016/j.carrev.2021.03.013. Epub 2021 Mar 20. PMID 33781677
- [Result] Louvard Y, Medina A. Definitions and classifications of bifurcation lesions and treatment. EuroIntervention. 2015;11 Suppl V:V23-6. doi: 10.4244/EIJV11SVA5. PMID 25983165

RESULTS

PARTICIPANT FLOW:
Groups:
- Scoreflex NC Scoring Percutaneous Transluminal Coronary Angioplasty (PTCA) Catheter: Single arm with investigational Scoreflex NC Scoring PTCA catheters
  Scoreflex NC Scoring PTCA catheter: To dilate coronary arteries during the subject's index procedure with Scoreflex NC Scoring PTCA catheters
Period: Overall Study
Arm/Group | Scoreflex NC Scoring Percutaneous Transluminal Coronary Angioplasty (PTCA) Catheter
Started | 200
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Lesions
Arm/Group | Scoreflex NC Scoring PTCA Catheter
Number analyzed (Participants) | 200
Number analyzed (Lesions) | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 154
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2
  Race: Black | 18
  Race: White | 178
  Race: Native Hawaiian/Pacific Islander | 1
  Race: American Indian/Alaska Native | 0
  Race: Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 200
Cardiac History [Count of Participants; unit: Participants] — More than one Cardiac History measure may be reported for each participant.
  Participants
    Prior Percutaneous Coronary Intervention | 106
    Prior Coronary Artery Bypass Graft | 26
    Prior Myocardial Infarction | 61
Current Cardiac Status [Count of Participants; unit: Participants]
  Asymptomatic | 18
  Silent Ischemia | 8
  Stable Angina | 116
  Unstable Angina | 57
  ST-Elevation Myocardial Infarction (STEMI) | 1
Cardiac Risk Factors [Count of Participants; unit: Participants] — More than one Cardiac Risk Factor may be reported for each participant.
  Participants
    Cigarette Smoking (within 30 days) | 37
    Diabetes Mellitus | 88
    Diabetes Mellitus (Insulin requiring) | 20
    Hypercholesterolemia Requiring Treatment | 181
    Hypertension Requiring Treatment | 182
Angiographic Characteristics: Vessel Location (Core Lab assessed) [Count of Units; unit: Lesions] — Analysis is based on the core lab assessed number of lesions (n=221).
  Lesions
    Left Anterior Descending Artery (LAD) | 97
    Left Circumflex Artery (LCX) | 55
    Right Coronary Artery (RCA) | 68
    Not Identified | 1
Angiographic Characteristics: Lesion Location (Core Lab assessed) [Count of Units; unit: Lesions] — Analysis is based on the core lab assessed anatomic position in the vessel. The total number of lesions assessed is 221.
  Lesions
    Ostial | 7
    Proximal | 98
    Middle | 93
    Distal | 23
Angiographic Characteristics: Lesion Characteristics (Core Lab assessed) [Mean (Standard Deviation); unit: Millimeters] — Analysis is based on the core lab assessed number of lesions (n=221).
  Millimeters
    Lesion Length | 18.37 (12.93)
    Minimal Luminal Diameter | 0.8 (0.40)
Angiographic Characteristics: Lesion Characteristics (Core Lab assessed) [Count of Units; unit: Lesions] — Analysis is based on the core lab assessed number of lesions (n=221).
  Lesions
    Moderate/Severe Calcification | 81
    Moderate/Severe Tortuosity | 7
    Total Occlusion | 11
Baseline Thrombolysis in Myocardial Infarction (TIMI) Flow (Core Lab assessed) [Count of Units; unit: Lesions] — Analysis is based on the core lab assessed number of lesions (n=221).
  Lesions
    0 (no perfusion) | 6
    1 (penetration with minimal perfusion) | 5
    2 (partial perfusion) | 6
    3 (complete perfusion) | 204
Angiographic Characteristics: Bifurcations, Medina Type (Core Lab assessed) [Count of Units; unit: Lesions] — The Medina Type is a classification system of the types of significant lesions in the 3 segments of a bifurcation as determined angiographically.
  A value of 0 or 1 (0 in the absence of significant stenosis and 1 in the presence of a stenosis >50%) is assigned to each of the 3 segments separated in the following order: proximal segment (PM), main distal segment (DM),side branch (SB), the values being separated by commas.(e.g. 1,1,1 would be considered the most complex with disease in all 3 segments.) Medina classification analysis results based upon all angiographic core lab lesions (n=221).
  Lesions
    0,0,0 | 2
    0,0,1 | 3
    0,1,0 | 38
    1,0,0 | 16
    0,1,1 | 8
    1,0,1 | 3
    1,1,0 | 8
    1,1,1 | 6
    Non-bifurcation lesions | 137

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device Procedural Success
Description: Device procedural success consisting of the following:
  * Successful delivery, inflation, deflation, and withdrawal of the study balloon
  * No evidence of vessel perforation, flow limiting dissection (grade C or higher) or reduction in Thrombolysis In Myocardial Infarction (TIMI) flow from baseline as related to the Scoreflex NC study balloon
  * Final TIMI flow grade of 3 at the conclusion of the percutaneous coronary intervention (PCI) procedure
Time Frame: Peri-procedural (at Day 0)
Population: Analysis population consists of intent-to-treat subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | Scoreflex NC Scoring PTCA Catheter
Number analyzed (Participants) | 200
Participants | 187

2. Secondary Outcome: Number of Participants With Angiographic Procedural Success
Description: Angiographic Procedural Success defined as Final diameter stenosis ≤ 50% in at least one of the Scoreflex NC attempted lesions following completion of the interventional procedure, including adjunctive stenting
Time Frame: Peri-procedural (at Day 0)
Population: Analysis population consists of intent-to-treat subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | Scoreflex NC Scoring PTCA Catheter
Number analyzed (Participants) | 200
Participants | 197

3. Secondary Outcome: Number of Participants With In-hospital Major Adverse Cardiac Events (MACE)
Description: In-hospital Major Adverse Cardiac Events (MACE), a composite of:
  * All death (cardiac and non-cardiac)
  * Myocardial infarction (MI)
  * Target Lesion Revascularization (TLR), clinically indicated
Time Frame: Endpoints will be measured through hospital discharge (expected to be within 24 hours)
Population: Analysis population consists of intent-to-treat subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | Scoreflex NC Scoring PTCA Catheter
Number analyzed (Participants) | 200
Participants | 9

4. Secondary Outcome: Number of Participants With In-hospital Stent Thrombosis (ST) Within the Target Vessel
Description: In-hospital stent thrombosis (ST) within the Target Vessel
Time Frame: Endpoint will be measured through hospital discharge (expected to be within 24 hours)
Population: Analysis population consists of intent-to-treat subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | Scoreflex NC Scoring PTCA Catheter
Number analyzed (Participants) | 200
Participants | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Arrhythmias (Requiring Intervention)
Description: Clinically Significant Arrhythmias (Requiring Intervention)
Time Frame: Endpoint will be measured through hospital discharge (expected to be within 24 hours)
Population: Analysis population consists of intent-to-treat subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | Scoreflex NC Scoring PTCA Catheter
Number analyzed (Participants) | 200
Participants | 1

6. Secondary Outcome: Number of Scoreflex NC Scoring Catheters That Had Occurrence of Balloon Rupture
Description: Occurrence of Scoreflex NC Study Balloon rupture
Time Frame: Peri-procedural
Population: Analysis population consists of intent-to-treat subject population. Site reported data represented on the use of 239 Scoreflex NC Scoring PTCA catheter study devices.
Measure: Count of Units; unit: Scoreflex NC Scoring PTCA catheters
Units Other Than Participants: Scoreflex NC Scoring PTCA catheters
Arm/Group | Scoreflex NC Scoring PTCA Catheter
Number analyzed (Participants) | 200
Number analyzed (Scoreflex NC Scoring PTCA catheters) | 239
Scoreflex NC Scoring PTCA catheters | 2

7. Secondary Outcome: Number of Participants That Had Improvement in Minimum Lumen Diameter (MLD) Following Use of Scoreflex NC Catheter (Measured by Quantitative Coronary Angiography (QCA))
Description: Improvement in Minimum Lumen Diameter (MLD) following use of Scoreflex NC catheter (measured by QCA).
  Improvement in MLD is defined as MLD post use of Scoreflex as greater than MLD from baseline.
Time Frame: Peri-procedural
Population: Analysis population consists of intent-to-treat subject population. Please note that the data for Number of Participants that had Improvement in Minimum Lumen Diameter was not analyzable in 23 patients by the Angiographic Core Lab.
Measure: Count of Participants; unit: Participants
Arm/Group | Scoreflex NC Scoring PTCA Catheter
Number analyzed (Participants) | 177
Participants | 161

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the point of subject enrollment through study completion at hospital discharge (hospital stay expected to be an average of 24 hours).
Arm/Group | Scoreflex NC Scoring PTCA Catheter
All-Cause Mortality (participants affected / at risk) | 0/200
Serious Adverse Events (participants affected / at risk) | 1/200
Other Adverse Events (participants affected / at risk) | 8/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scoreflex NC Scoring PTCA Catheter (N=200)
Target Lesion Revascularization Clinically Indicated TLR) (Cardiac disorders) | 1 (1)
Myocardial Infarction (Non Q-wave) (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scoreflex NC Scoring PTCA Catheter (N=200)
Myocardial Infarction (Non Q-wave) (Cardiac disorders) | 7 (7)
Clinically Significant Arrhythmias (Requiring Intervention) (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT03763747/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT03763747/SAP_001.pdf